CLINICAL TRIAL: NCT01688726
Title: Evaluation of SYSTANE® BALANCE on Conjunctival Staining (CS) Visual Performance (VP) and Tear Film Kinetics (TFK) in Dry Eye Subjects With Lipid Deficiency
Brief Title: Evaluation of SYSTANE® BALANCE in Dry Eye Subjects With Lipid Deficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A00977
Record Dates: First submitted 2012-09-17; First posted 2012-09-20 (Estimated); Results first posted 2014-11-18 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2014-08

CONDITIONS: Dry Eye Syndrome; Lipid Deficiency
Keywords: Dry eye; Ocular surface; Vision complaint; Tear film stability; Time controlled functional visual acuity; Tear film kinetics
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SYSTANE BALANCE (Experimental): SYSTANE® BALANCE eyedrops, 1 drop 4 times a day for a continuous period of 1 month
  Interventions: Other: SYSTANE® BALANCE eyedrops
- Minims Saline (Active Comparator): Minims® Saline 0.9% eyedrops, 1 drop 4 times a day for a continuous period of 1 month
  Interventions: Other: Minims® Saline 0.9% eyedrops

INTERVENTIONS:
Other: SYSTANE® BALANCE eyedrops
  Arms: SYSTANE BALANCE
Other: Minims® Saline 0.9% eyedrops
  Arms: Minims Saline

SUMMARY:
The purpose of this study is to evaluate the repeated use of SYSTANE® BALANCE on stabilizing the tear film of dry eye patients with an unstable tear film.

ELIGIBILITY:
Inclusion Criteria:

* Non-contact lens wearer;
* Symptomatology as defined by the Ocular Surface Disease Index (OSDI) questionnaire;
* Lipid deficiency;
* Best visual acuity of 6/9 or better in each eye;
* Willingness to adhere to the instructions set in the clinical protocol;
* Signature of the subject informed consent form;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Use of systemic medication which might produce dry eye side effects;
* Systemic disease which might produce dry eye side effects;
* Active or recent ocular inflammation or infection;
* Use of ocular medication;
* Significant ocular anomaly;
* Previous ocular surgery;
* Previous use of Restasis;
* Any medical condition that might be prejudicial to the study;
* Pregnant or lactating;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2012-12; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michel Guillon, PhD, FCOptom, FAAO, CCTI, Principal Investigator — OTG Research & Consultancy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 1 clinical site located in the UK.
Pre-assignment Details: A total of 91 participants were enrolled and randomized. This reporting group includes all randomized participants (91).
Groups:
- SYSTANE BALANCE; Minims Saline: One drop 4 times a day for a continuous period of 1 month
Period: Overall Study
Arm/Group | SYSTANE BALANCE | Minims Saline
Started | 46 | 45
Completed | 45 | 44
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Relocated abroad | 0 | 1

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | SYSTANE BALANCE | Minims Saline | Total
Number analyzed (Participants) | 46 | 45 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (16.51) | 44.6 (14.84) | 45.7 (15.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 29 | 59
  Male | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Mean Bulbar Conjunctival Staining
Description: The conjunctival staining present in the bulbar area was evaluated 120 minutes post eyedrop instillation using a slit lamp with digital image capture and lissamine green strips. Staining coverage as a percentage of the exposed bulbar conjunctiva is reported. A lower percentage in staining area represents a better outcome.
Time Frame: Month 1
Population: This analysis population includes all randomized participants with at least 1 evaluable post-treatment efficacy assessment.
Measure: Mean (Standard Deviation); unit: percentage of staining
Arm/Group | SYSTANE BALANCE | Minims Saline
Number analyzed (Participants) | 45 | 44
percentage of staining
  Right eye | 0.743 (1.685) | 0.442 (0.999)
  Left eye | 0.531 (1.056) | 0.443 (1.404)

2. Secondary Outcome: High Contrast logMAR Time Controlled Visual Acuity (TCVA)
Description: TCVA (functional visual performance) was measured with both eyes together under controlled lighting, contrast and temporal conditions using the OTG computerized vision testing system prior to eyedrop instillation (baseline) and at 60, 90, and 120 minutes post eyedrop instillation with the subject's up-to-date vision correction in place. TCVA is measured in logarithm of the minimum angle of resolution (logMAR), with logMAR acuity of 0.0 considered normal distance eyesight. A negative logMAR value denotes better visual acuity.
Time Frame: Month 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | SYSTANE BALANCE | Minims Saline
Number analyzed (Participants) | 45 | 44
logMAR
  Baseline | 0.220 (1.105) | 0.253 (0.100)
  60 minutes | 0.206 (1.106) | 0.295 (0.840)
  90 minutes | 0.240 (1.124) | 0.202 (0.826)
  120 minutes | 0.293 (1.090) | 0.206 (0.973)

3. Secondary Outcome: Non Invasive Tear Film Break-up-time (NIBUT)
Description: NIBUT was measured prior to eyedrop instillation (baseline) and at 60, 90, and 120 minutes post eyedrop instillation. The time elapsed between eye opening after a blink and the appearance of the first dark spot within the tear film as observed with a specialized illumination source was recorded. A higher number represents a lengthening in the tear film break up time and greater perceived ocular comfort.
Time Frame: Month 1
Population: This analysis population includes all randomized participants with at least 1 evaluable post-treatment efficacy assessment. Here, n represents the number of participants with non-missing values at the specific time point for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- SYSTANE BALANCE/Right Eye; SYSTANE BALANCE/Left Eye; Minims Saline/Right Eye; Minims Saline/Left Eye: One drop 4 times a day for 1 month
Arm/Group | SYSTANE BALANCE/Right Eye | SYSTANE BALANCE/Left Eye | Minims Saline/Right Eye | Minims Saline/Left Eye
Number analyzed (Participants) | 45 | 45 | 44 | 44
seconds
  Baseline (n=44,44) | 9.39 (7.68) | 7.47 (7.38) | 9.53 (13.19) | 7.66 (8.32)
  60 minutes (n=44,43) | 7.81 (10.17) | 8.74 (10.42) | 8.17 (10.45) | 6.96 (6.16)
  90 minutes (n=44,43) | 8.41 (9.55) | 7.59 (9.64) | 7.31 (8.33) | 6.97 (5.39)
  120 minutes (n=44,43) | 6.92 (6.52) | 7.26 (6.71) | 8.63 (10.08) | 6.16 (6.59)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study (Dec2012 to Nov2013). This analysis population includes all subjects who were randomized into the study, used at least 1 eye drop, and completed at least 1 post-treatment safety assessment.
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the medical device.
Arm/Group | SYSTANE BALANCE | Minims Saline
Serious Adverse Events (participants affected / at risk) | 1/46 | 1/45
Other Adverse Events (participants affected / at risk) | 0/46 | 0/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SYSTANE BALANCE (N=46) | Minims Saline (N=45)
Blood poisoning (Infections and infestations) | 1 | 0
Knee operation (Surgical and medical procedures) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.